CLINICAL TRIAL: NCT01566448
Title: Treatment of Severe Mucositis Pain With Oral Ketamine Mouthwash
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aaron Cumpston, PharmD, BCOP (Other)
Responsible Party: Sponsor-Investigator, Aaron Cumpston, PharmD, BCOP, Pharmacy Clinical Specialist (Principal Investigator), West Virginia University
Organization: West Virginia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVU041011
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Mucositis
Keywords: Ketamine; Mucositis; Oral ketamine rinse
MeSH Terms: conditions — Mucositis | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketamine (Experimental): Ketamine oral mouthwash 20mg/5ml swish and spit four times daily
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 20mg/5ml swish and spit four times daily

SUMMARY:
Oral mucositis (inflammation of the lining of the mouth) is a very common adverse effect when chemotherapy and radiation therapy are used to treat cancer. Mucositis occurs in about 40% of patients receiving standard dose chemotherapy, 80% of patients receiving radiation therapy of the head and neck, and up to 100% of patients undergoing a bone marrow transplant. Because the pain from mucositis can be so bad it can cause the inability to eat or drink, inability to talk, gagging and drooling. Many times mucositis can affect cancer treatment because patients may have to be given a lower dose of a drug or stop treatment completely. There are not many treatments today that can help relieve the severe pain caused from mucositis. This research study will help researchers determine if using an oral mouthwash called Ketamine will help lessen mucositis pain.

Ketamine is approved by the Food and Drug Administration (FDA) for use with general anesthesia, sedation and for severe pain. WVU Hospital is now using Ketamine mouthwash as a standard treatment option for mucositis pain.

During this study patients will be assessed to determine the level of pain caused by their mucositis. This will occur before the first dose, one hour after the first dose, and then daily until they are no longer on the study. Patients will use the mouthwash by swishing and spitting (20mg/5ml) four times each day, and also every four hours as needed. Patients will use the mouthwash on this study until their mucositis gets better or until the mucositis gets worse (or if the pain does not get better after three days of treatment).

DETAILED DESCRIPTION:
Mucositis

Mucositis is an adverse effect as a result of chemotherapy and radiation treatments and has significant quality of life and clinical consequences. Mucositis is a result of direct cytotoxic damage as well as a cytokine-mediated inflammatory response and can affect the epithelial mucosal surfaces along the entire gastrointestinal tract. Mucositis manifesting in the oral cavity can be especially distressing to patients and may involve erythema, cracking, inflammation, bleeding and ulceration and typically begins 5-10 days after starting chemotherapy. Mucositis occurs in about 40% of patients receiving standard dose chemotherapy, 80% of patients receiving radiation therapy to the head and neck, and up to 100% of patients undergoing a bone marrow transplant.(1)

Pain from oral mucositis has been reported as the single most debilitating side effect by patients receiving bone marrow transplants. Mucositis is also the most common condition requiring analgesics during cancer therapy. Complications of pain from mucositis include inability to tolerate food or fluid intake, difficulty or inability to talk, excess mucus, gagging, sleep disturbances, and drooling. Mucositis may also require hospital admission or extended admission for total parenteral nutrition, intravenous analgesia, and/or intravenous antibiotics. Seventy percent of patients with a grade 3 or 4 mucositis will require a feeding tube. Mucositis also has the potential to impact the effectiveness of cancer treatment as it is a dose-limiting toxicity and results in cessation or reduction of treatment in 35% of patients (2,3,4)

Current standard of care focuses on palliation and includes systemic opiate analgesics for moderate to severe mucositis pain, topical anesthetics and mucosal coating agents such as lidocaine, benzocaine, dyclonine, diphenhydramine, doxepin, and benzydamine for moderate pain, and bland rinses for mild pain. Data supporting these management options are limited. Other agents that have been investigated with variable responses are oral capsaicin, oral sulfasalazine, and growth factor mouthwashes. (5)

Ketamine

Ketamine is a sedative hypnotic with anesthetic and analgesic properties. Ketamine works by selectively depressing the thalamoneocortical system, non-competitively blocking N-methyl-D-aspartate (NMDA) receptors, and having intrinsic sympathomimetic activity. Ketamine also appears to selectively interrupt association pathways in the brain producing somatesthetic sensory blockade. Ketamine is FDA-approved for induction and maintenance of general anesthesia but has also been used for procedural sedation, refractory severe pain, and acute respiratory failure in children. (6)

Topical administration of ketamine was shown to cause a reduction in allodynia in a double-blind placebo controlled study and peripheral administration of ketamine has antinociceptive efficacy similar to that of systemic administration which is likely mediated by NMDA antagonism (7). Ketamine may also potentiate the effects of other systemic opioid analgesics and may reverse opiate tolerance to some degree. Also, given that topical administration of opiates has a local effect, topical ketamine may produce a local tolerance reversal. Ketamine also has modest anti-inflammatory properties which could provide beneficial effects in mucositis pain relief. (8)

Ketamine oral rinse use was described in a case report of a 32 year old female with radiation-induced mucositis pain refractory to Clark's solution, transdermal fentanyl, and intravenous hydromorphone. Ketamine oral rinse was given as 20mg of drug in a 5ml artificial saliva solution every 3 hours as needed with continued PCA use. She experienced decreased pain at rest and with eating and was able to decrease the dose of her opiate analgesics. Her overall pain was reported as decreased from 9/10 to 3/10 with oral ketamine use. No adverse effects were reported other than one episode of swallowing the solution which resulted in transient sedative and psychomotor effects. (8)

A retrospective chart review of ketamine mouthwash use in 8 patients over a period of 4 years was conducted to determine safety and efficacy. Patients in this review received ketamine 20mg/5ml mouthwashes every 4 hours as needed. Seven of the 8 patients were post-hematopoietic stem cell transplant (post-HSCT) patients. Five patients had a documented improvement in mucositis pain and 4 patients experienced an adverse event. Adverse events consisted of mild confusion, nausea, vertigo, and hallucinations; however 2 of the 4 patients had reports of these symptoms prior to beginning ketamine mouthwashes but were still included in the analysis. Patients received an average of 17 doses over an average of 6 days. Reporting of pain scores were variable and difficult to quantify but the authors concluded that ketamine may provide a viable treatment option for mucositis pain. (9)

Rationale for study

Evidence for the use of an oral ketamine rinse suggests that it could provide a distinct benefit for patients suffering from pain and other clinical consequences of mucositis as a result of cancer treatments. No treatment is currently available that provides a profound relief from this pain and available evidence suggests that ketamine could be a useful tool in the arsenal of agents available to patients. Ketamine mouthwash was approved by the WVUH Pharmacy Nutrition and Therapeutics (PNT) Committee as a treatment option for mucositis pain. It is commercially available and currently used at our hospital. No prospective data exists objectively evaluating the potential benefits and possible adverse effects of ketamine oral rinse. We postulate that using ketamine as an oral mouthwash will provide pain relief for patients with significant distress due to pain from oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Patient has oral mucositis pain that is grade 3 or 4 according to the World Health Organization (WHO) Oral Mucositis Scale
* Patient has received at least one prior chemotherapy or radiation treatment
* Patient is at least 18 years old
* Patient or their legally authorized representative understands and voluntarily signs the written informed consent prior to any study-specific procedures. A copy of the signed informed consent form will be retained by the treating institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Cumpston, PharmD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospitals Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

REFERENCES:
- [Background] Harris DJ. Cancer treatment-induced mucositis pain: strategies for assessment and management. Ther Clin Risk Manag. 2006 Sep;2(3):251-8. doi: 10.2147/tcrm.2006.2.3.251. PMID 18360600
- [Background] Bellm LA, Epstein JB, Rose-Ped A, Martin P, Fuchs HJ. Patient reports of complications of bone marrow transplantation. Support Care Cancer. 2000 Jan;8(1):33-9. doi: 10.1007/s005209900095. PMID 10650895
- [Background] Sonis ST, Elting LS, Keefe D, Peterson DE, Schubert M, Hauer-Jensen M, Bekele BN, Raber-Durlacher J, Donnelly JP, Rubenstein EB; Mucositis Study Section of the Multinational Association for Supportive Care in Cancer; International Society for Oral Oncology. Perspectives on cancer therapy-induced mucosal injury: pathogenesis, measurement, epidemiology, and consequences for patients. Cancer. 2004 May 1;100(9 Suppl):1995-2025. doi: 10.1002/cncr.20162. PMID 15108222
- [Background] Borbasi S, Cameron K, Quested B, Olver I, To B, Evans D. More than a sore mouth: patients' experience of oral mucositis. Oncol Nurs Forum. 2002 Aug;29(7):1051-7. doi: 10.1188/02.ONF.1051-1057. PMID 12183754
- [Background] Bensinger W, Schubert M, Ang KK, Brizel D, Brown E, Eilers JG, Elting L, Mittal BB, Schattner MA, Spielberger R, Treister NS, Trotti AM 3rd. NCCN Task Force Report. prevention and management of mucositis in cancer care. J Natl Compr Canc Netw. 2008 Jan;6 Suppl 1:S1-21; quiz S22-4. PMID 18289497
- [Background] Ketamine. Clinical Pharmacology Online. Elsevier/Gold Standard, Inc. 15 Nov 2011.
- [Background] Finch PM, Knudsen L, Drummond PD. Reduction of allodynia in patients with complex regional pain syndrome: A double-blind placebo-controlled trial of topical ketamine. Pain. 2009 Nov;146(1-2):18-25. doi: 10.1016/j.pain.2009.05.017. Epub 2009 Aug 22. PMID 19703730
- [Background] Slatkin NE, Rhiner M. Topical ketamine in the treatment of mucositis pain. Pain Med. 2003 Sep;4(3):298-303. doi: 10.1046/j.1526-4637.2003.03032.x. PMID 12974832
- [Background] Ryan AJ, Lin F, Atayee RS. Ketamine mouthwash for mucositis pain. J Palliat Med. 2009 Nov;12(11):989-91. doi: 10.1089/jpm.2009.0198. PMID 19708855
- [Derived] Shillingburg A, Kanate AS, Hamadani M, Wen S, Craig M, Cumpston A. Treatment of severe mucositis pain with oral ketamine mouthwash. Support Care Cancer. 2017 Jul;25(7):2215-2219. doi: 10.1007/s00520-017-3627-6. Epub 2017 Feb 11. PMID 28190158
- See also: West Virginia University Mary Babb Randolph Cancer Center — http://wvucancer.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Scores
Description: Change in pain score as reported at baseline and after the use of ketamine mouthwash on a numeric scale from 0 to 10, with 0 representing no pain and 10 representing the worst pain.
Time Frame: 1 hour after baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 30
score on a scale | 2 [0 to 10]

2. Secondary Outcome: Time From Dose Administration to Change in Pain Intensity as Reported by Subject.
Description: Patients will be questioned about time until maximal pain relief and given options of: no effect, 1-15 minutes, 15-30 minutes, 30-45 minutes, 45-60 minutes and greater than 1 hour.
Time Frame: 1 day after start of ketamine mouthwashes
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine
Number analyzed (Participants) | 30
Participants
  No effect | 2
  0-15 minutes | 28

3. Secondary Outcome: Duration of Effect of Pain Reduction
Description: Patients will be question about the duration of pain relief and given the option of no effect, less than one hour, 1-2 hours, 2-3 hours, 3-4 hours, greater than 4 hours or N/A.
Time Frame: Day 1 after start of ketamine mouthwashes
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine
Number analyzed (Participants) | 30
Participants
  <1 hour | 14
  1-2 hours | 7
  2-3 hours | 6
  3-4 hours | 0
  >4 hours | 1
  No effect | 2

4. Secondary Outcome: Change in Use of Narcotic Analgesics
Description: Change in IV morphine equivalents of opioid requirements
Time Frame: Days 1 after start of ketamine mouthwashes
Measure: Median (Full Range); unit: IV morphine equivalents
Arm/Group | Ketamine
Number analyzed (Participants) | 30
IV morphine equivalents | 12 [0 to 202]

5. Secondary Outcome: Change in Topical Lidocaine Usage
Description: Change of topical lidocaine uses in 24 hour period
Time Frame: Days 1 after start of ketamine mouthwashes
Measure: Median (Full Range); unit: lidocaine doses per day
Arm/Group | Ketamine
Number analyzed (Participants) | 30
lidocaine doses per day | 1 [0 to 8]

6. Secondary Outcome: Change in Sleep Quality
Description: Sleep quality, as reported by the subject on a numeric scale (1-10) will be used as a surrogate marker of quality of life with 0 indicating no sleep and 10 indicating the best sleep you have had.
Time Frame: Day 1 after start of ketamine mouthwashes
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 30
score on a scale | 1 [1 to 10]

ADVERSE EVENTS:
Arm/Group | Ketamine
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes